CLINICAL TRIAL: NCT04420065
Title: CompaRative Study of the Effects of Left ventriculAr and Biventricular Pacing on inDices of cArdiac Function and Clinical Course of Heart Failure PatienTs: Rationale and Design of the READAPT Randomized Trial
Brief Title: Effects of Preferential Left Ventricular Pacing on Ventriculoarterial Coupling and Clinical Course of Heart Failure
Acronym: READAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Christina Chrysohoou, Cardiology Consultant, Director of Cardiology, Senior Researcher, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: READAPT
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart failure; Cardiac resynchronization therapy; Preferential left ventricular pacing; Ventriculoarterial coupling; Echocardiography; Cardiopulmonary exercise test
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: Patients randomized after enrollment to receive either standard biventricular pacing, or preferential left ventricular pacing (left ventricle will be resynchronized, but right ventricle will be activated through the intrinsic conduction system)
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and assessor unaware of chosen programming mode and activated algorithms. The standard of care that is biventricular pacing will be provided to all participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Classical biventricular pacing (Active Comparator): Commercially available LV-pacing capable CRT devices and quadripolar leads will be implanted. Right ventricular (RV) and right atrial (RA) leads will be placed according to standard practice. The LV lead will also be placed according to standard practice, targeting to a lateral, posterolateral, or anterolateral branch of the coronary sinus (CS). Interventricular delay programmed will be determined based on stroke volume maximization, and will be used as a criterion for BVP optimization. Atrioventricular delay optimization shall be automatically performed by the device.
  Interventions: Device: Biventricular pacing
- Preferential left ventricular pacing (Experimental): In G2 patients, an algorithm for preferential left ventricular pacing will be activated. Following selection of the dipole maximizing stroke volume during simultaneous LV-RV pacing, subsequent V-V delay optimization shall be delegated to the algorithm. Based on previous studies, a subgroup analysis of G2 will be performed, comparing those receiving ≥50% with those receiving <50% preferential LV pacing evaluated over the total duration of the study (12 months).
  Interventions: Device: Preferential left ventricular pacing

INTERVENTIONS:
Device: Preferential left ventricular pacing — Activation of an algorithm attempting to provide preferential left ventricular pacing in an anticipatory manner, thus potentially preventing iatrogenic, pacing-related, right ventricular dysfunction, and improving coupling and outcomes in dyssynchronous heart failure patients
  Arms: Preferential left ventricular pacing
Device: Biventricular pacing — Standard biventricular pacing, with V-V delay programmed based on stroke volume maximization, and A-V delay delegated to the device
  Arms: Classical biventricular pacing

SUMMARY:
Randomized trial of adult patients to study the effects of preferential left ventricular pacing on ventriculoarterial coupling of both systemic and pulmonary circulation, indices of systolic and diastolic function of both ventricles, and clinical course of patients with advances dyssynchronous heart failure.

DETAILED DESCRIPTION:
Study hypothesis is that preferential left ventricular (LV) pacing, delivered by means of the AdaptivCRT® algorithm and in conjunction with automated V-V delay adjustments, will lead to improvements over standard biventricular pacing (BVP) in the function of all cardiac chambers, reduce arrhythmic burden, improve ventricular-arterial coupling (VAC), and patient functional status. It would be interesting to study what changes in right-side VAC (RVAC) can be appreciated with the activation of the preferential LV pacing algorithm and how they relate to each other, i.e. whether LV is driven towards maximizing output whilst RV shifts to optimizing energy efficiency.

READAPT is a single-center, prospective, randomized trial of heart failure patients eligible for CRT according to current European heart failure guidelines. Informed written consent is required from all study participants.

Adult (aged 18-80 years old), consenting patients with any cardiomyopathy type, diagnosed at least 6 months prior (to exclude recent myocarditis cases that may remit and confound outcomes), on optimal medical therapy for at least 3 months, and an existing I/IIa indication for a cardiac resynchronization therapy - defibrillator (CRT-D) device will be enrolled and randomized into 2 groups, one receiving standard CRT (Group 1 - G1), and one with activation of the preferential LV pacing algorithm (Group 2 - G2). Enrollment date will amount to the baseline assessment date, with device implantation occurring preferably within 48 hours. READAPT will include patients with both new CRT-D implantation and an upgrade from an existing defibrillator or pacemaker with no prior left ventricular lead placement.

ELIGIBILITY:
Inclusion Criteria:

Age 18-80 years old Provided informed consent Any cardiomyopathy type, diagnosed at least 6 months prior (to exclude recent myocarditis cases that may remit and confound outcomes) On optimal medical therapy for at least 3 months, An existing I/IIa indication for a CRT-D device Both new CRT-D implantation and an upgrade from an existing ICD or pacemaker with no prior left ventricular lead placement.

Exclusion Criteria:

1. Have an existing Class I recalled lead,
2. Are anticipated to need heart transplantation within the next 9 months,
3. Have undergone cardiac transplantation less than 40 days prior to enrolment,
4. Have had a cerebrovascular accident or transient ischemic attack within 3 months of enrollment,
5. Have had a recent myocardial infarction less than 40 days prior to enrollment, or unstable angina or cardiac revascularization less than 3 months prior to enrolment,
6. Have documented moderate to severe/severe mitral/aortic/tricuspid/pulmonary insufficiency (noninvasive VAC calculation impossible),
7. Exhibit a daily burden of premature ventricular complexes (PVCs) of either ≥10% of total QRSs or ≥10,000 on ambulatory ECG recording21, 22 (to exclude PVC-related, potentially reversible cardiomyopathy),
8. Are currently participating in a clinical investigation that includes an active treatment arm,
9. Have diagnosed pulmonary hypertension other than class II (left heart-related),
10. Have known stage IV-V renal dysfunction (clearance estimated by the Cockcroft-Gault equation),
11. Have permanent atrial fibrillation,
12. Have complete atrioventricular block,
13. Have a prolonged (>200msec) PQ interval on surface ECG (thus invalidating the option for preferential LV pacing),
14. Are pregnant or planning to become pregnant during the duration of the study (in case of unplanned pregnancy the patient will have to be excluded from the study),
15. Have an expected life expectancy of <12 months, or
16. Undergo major adaptations to their pharmacological regimens during follow-up (e.g. initiation of neprilysin inhibitors).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in patient exercise capacity | 12 months
  Assessed by cardiopulmonary exercise test in terms of maximal oxygen consumption in ml/kg/min

SECONDARY OUTCOMES:
Number of hospitalizations for heart failure | 12 months
  Data retrieved from online patient file will be used to compare number of unplanned hospitalizations for worsening heart failure between groups
Left ventricular function | 12 months
  Assessed by ejection fraction (in %), strain echocardiography - changes in % global longitudinal peak strain and diastolic function indices (E/e')
Right ventricular function | 12 months
  Assessed by strain echocardiography in terms of two-dimensional % global longitudinal peak strain
Ventriculoarterial coupling for both systemic and pulmonary circulation | 12 months
  Assessed by the noninvasive single-beat echocardiographic method in terms of distance from 1 (value associated with maximization of stroke work for a given contractility)

CONTACTS AND LOCATIONS:
Locations (1):
- First University Department of Cardiology, Hippokrateion General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Study design data and anonymized individual data allowing for pooling in subsequent analyses
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data to be shared 2 years after study completion
Access Criteria: Request made by investigator with an active, registered clinical trial